CLINICAL TRIAL: NCT00453011
Title: CSP #338 - Comparison of Anterior and Posterior Chamber Lens Implants After Vitreous Loss in Attempted Extracapsular Cataract Extraction
Brief Title: Comparison of AC and PC Lenses After Vitreous Loss During ECCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 338
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Cataract
Keywords: vitreous loss; intraocular lenses; Patients undergoing extracapsular cataract surgery; Vitreous loss with sufficient capsular support for an unsutured posterior chamber lens; 5% random sample of patients with no vitreous loss
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Device: posterior chamber intraocular lens
Device: anterior chamber intraocular lens

SUMMARY:
Objective: The standard definition of failure in cataract surgery is best corrected visual acuity of less than 20/40 at one year. The specific aim of this cooperative study was to compare the failure rate for those patients with vitreous loss in whom an PC IOL is placed to the failure rate for those in whom an AC IOL is placed after vitreous loss.

Design: A total of 437 patients in 15 centers were randomized to AC or PC IOL over a 45-month period and were followed for a minimum of one year. The null hypothesis is that the rate of failure is the same in the two groups.

All patients who were about to undergo cataract surgery in the participating centers and who did not meet an exclusion criterion were eligible for the study. At the time of surgery, if there was vitreous loss, and if in the opinion of the surgeon there was sufficient capsular support for a posterior chamber lens to be placed, then the patient was randomized into one of either the anterior or posterior chamber lens groups. The patients were then followed for complications (e.g., retinal detachment, cystoid macular edema, uveitis, glaucoma, hyphema) and for the primary end point of visual acuity of 20/40 or better at one postoperative year.

An "Index Group" of about 500 patients without vitreous loss also were followed according to study protocol. These patients were compared to those in the PC and AC IOL groups with respect to outcome and baseline characteristics in order to assess the effect of vitreous loss on complication rates.

All patients were followed at annual intervals until the termination of the study. This allowed the study to obtain long-term information with regard to visual acuity and complication rates.

DETAILED DESCRIPTION:
Primary Hypothesis: There is no difference in failure rate between patients receiving anterior chamber or posterior chamber intraocular lenses following vitreous loss in extracapsular cataract extraction (ECCE).

Secondary Hypothesis: None

Intervention: 1) Anterior chamber intraocular lens, 2) Posterior chamber intraocular lens.

Primary Outcome: Failure defined as best corrected visual acuity less than 20/40 one year following ECCE.

Study Abstract: Extracapsular cataract surgery with posterior chamber intraocular lens implantation is one of the most common and most successful of surgical procedures. In the United States alone approximately 1.4 million cataract extractions were performed in 1990. Of these the overwhelming majority do well. However, the principal complication, vitreous loss, occurs in about 5% of cases. It is often sight-limiting.

Placement of an intraocular lens in the presence of vitreous loss is controversial. The standard approach following anterior vitrectomy usually involves placement of an anterior chamber intraocular lens (AC IOL). However, it has been suggested that implantation of a posterior chamber intraocular lens (PC IOL) in many of these patients is not only possible, but preferable.

In this study, eligible patients were VA patients who had vitreous loss during attempted ECCE. At each occurrence of vitreous loss, the patients were randomly assigned to have an AC IOL or PC IOL. Patient recruitment was terminated early with 438 patients enrolled in 15 centers. Patients were followed to the completion of at least one-year follow-up.

An ?Index Group?of 500 patients without vitreous loss also was followed according to study protocol. These patients will be compared to those in the PC and AC IOL groups with respect to outcome and baseline characteristics in order to assess the effect of vitreous loss on complication rates.

Results: More PC IOL patients (91%) achieved visual acuity of 20/40 or better at one year than AC IOL patients (79%). A highly significant difference (p=0.003). There was no significant difference between the two groups for patients' rating of vison or adverse events. Over 84% of the PC IOL patients and over 77% of the AC IOL patients rated their vision as good or better at one year as opposed to only 7% giving such ratings prior to surgery. For at least one rating period during the first year, 13.2% of the combined study patients had cystoid macular edema, 8.5% had posterior capsule opacification, 5.7% had glaucoma, and 3.7% had retinal detachment.

Conclusion: In the presence of sufficient capsular support, a PC IOL should be implanted after vitreous presentation during ECCE.

Collins JF, Krol WF, Gaster RN, Colling CL, Kirk GF, Smith TJ - A Comparison of Anterior Chamber and Posterior Chamber IOL's after Vitreous Loss during Cataract Surgery. The VA Cooperative Cataract Study. American Journal of Ophthalmology. 136:1-9, 2003

Collins JF, Krol WF, Kirk GF, Gaster, RN - The Effect of Vitreous Presentation During Extracapsular Cataract Surgery on the Postoperative Visual Acuity at One Year. American Journal of Ophthalmology. 138:536-542, 2004

Collins, JF, Gaster,RN, Krol,WF and the VA Cooperative Cataract Study Group. Outcomes in Patients Having Vitreous Presentation During Cataract Surgery Who Lack Capsular Support for a Nonsutured PC IOL. American Journal of Ophthalmology, Vol 141:71-78, 2006

ELIGIBILITY:
Inclusion Criteria:

* The principal eligibility criterion was a visually significant lens opacity resulting in a best-corrected distance visual acuity of 20/50 or worse.

Exclusion Criteria:

* Age less than 18 years
* Unwillingness to give informed consent
* Unwillingness to agree to protocol follow-up
* Visual acuity better than 20/50
* Any other ocular disease which would preclude a final postoperative visual acuity of 20/40 or better (e.g., proliferative diabetic retinopathy, flaucoma, or Fuchs' dystrophy)
* History of uveitis
* Other contraindication to an IOL
* Cataract attributable to trauma
* Patient only had one eye with potential for useful vision
* Any retinal thickening or definite hard exudates within one disk diameter of center of macula
* Patient's other eye already entered into the study.

Patients could be screened for the study twice; once for each eye if they had a cataract in both. However, if the first procedure resulted in the patient being entered into the randomized study, the 5% NVP group, or the ICS group, then the second eye was not eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202
Dates: Start 1992-02; Study Completion 1998-02

REFERENCES:
- [Derived] Gaster RN, Collins JF. The long-term effect of vitreous presentation during extracapsular cataract surgery on postoperative visual acuity. Am J Ophthalmol. 2007 Aug;144(2):186-194. doi: 10.1016/j.ajo.2007.04.023. Epub 2007 Jun 7. PMID 17559787